CLINICAL TRIAL: NCT04917601
Title: A Randomized Controlled Multicenter Study for Evaluating a Digital Support System in Childhood Obesity Treatment (EurEvira)
Brief Title: A Multicenter Study for Evaluating a Digital Support System in Childhood Obesity Treatment
Acronym: EurEvira
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Lund University (Other); Evira AB (Industry)
Responsible Party: Principal Investigator, Pernilla Danielsson, Pediatric nurse, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-05513; 2019-05513 (Other Grant/Funding Number: Vinnova)
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Childhood Obesity; Adolescent Obesity; mHealth; Personalized Medicine
Keywords: Obesity treatment; Digital support system
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Children aged 4-17 years old with obesity will be randomized to either the intervention group or the control group. The intervention group will through daily weighings at home be able to follow treatment closely in an application on the parents phone. Through a communication function in the application, families will be able to communicate in a fast and easy way with healthcare professionals at the clinic. The control group will receive Standard Lifestyle Care following local routines. The study duration is 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evira Care treatment (Experimental): The intervention arm will receive Evira Care in combination with Standard Lifestyle Care. If the standard treatment, after the first month of treatment, contains more frequent visits than every third month, the number of standard visits shall be reduced to a maximum of one visit every third month. During the first 2-4 weeks, participants will receive information about the system and how to utilize the daily weighings and communication system. The families will be informed about possible lifestyle changes that may be effective and that they are supposed to do lifestyle changes primarily regarding energy intake that they do consider feasible in their specific living situations.
  Clinical investigations will be completed and includes physical and abdominal examinations, weight, height, and blood pressure. All participants will also be asked to answer questionnaires including quality of life, eating disorders, and treatment satisfaction.
  Interventions: Behavioral: Evira Care treatment
- Standard Lifestyle Care (Active Comparator): The control group will receive the standard care of treatment for childhood obesity, which addresses lifestyles without any restriction in visits or clinical support.
  Clinical investigations will be completed and includes physical and abdominal examinations, weight, height, and blood pressure. All participants will also be asked to answer questionnaires including quality of life, eating disorders, and treatment satisfaction.
  Interventions: Behavioral: Standard Lifestyle Care

INTERVENTIONS:
Behavioral: Evira Care treatment — The intervention aim to examine the effectiveness of using a digital support system (Evira) in treatment of childhood obesity. Through daily weighings at home using a special designed scale, which sends data directly to an application on the parents phone and to a clinic homepage, the child's weight development can be easily monitored. Participants can be randomized to either the intervention group or the control group. The control group will receive local standard treatment.
  Arms: Evira Care treatment
Behavioral: Standard Lifestyle Care — The control group will receive the local standard care of treatment addressing lifestyles for childhood obesity without any restriction in visits or clinical support. This is the current standard care of treatment for childhood obesity.
  Arms: Standard Lifestyle Care

SUMMARY:
Evira is a digital support system newly developed for treatment of childhood obesity. Through daily weighings at home using a special scale together with a message function in the Evira application, enabling fast and easy communication with the clinic, parents and the clinicians can easily follow the child's weight development. The purpose of this randomized controlled study is to evaluate the effect of adding Evira to the already locally used life-style treatment of childhood obesity.

DETAILED DESCRIPTION:
Obesity in childhood is a global public health problem which continues to increase. It is associated with type 2 diabetes, high blood pressure, certain types of cancer, decreased psychosocial health and early mortality, among many other short- and long-term consequences. It is estimated that families of children with obesity need at least 26 hours of contact with the health care per year to make it possible for the children to reach a clinically relevant reduction in degree of obesity. Such visit frequency is difficult to carry out due to its cost for society and places great demands on families.

A digital support system named Evira has newly been developed and is based on four cornerstones; a) daily self-monitoring of weight, b) a mobile app used by parents to easily follow weight development, c) a website on which clinicians view the same data as parents do and d) communication between clinicians and parents by text messages through the website and the mobile app. Hence, Evira enables close follow-up of treatment results and continuous communication between the healthcare and the families.

The overall aim is to evaluate the effects of adding Evira, a digital support system for childhood obesity treatment and accompanying treatment manual, to the already locally used life-style treatment.

Boys and girls aged 4-17 years old with obesity will be asked for participation. All patient who fulfills the inclusion criteria and have signed the informed consent form will be included and randomized into the study. Randomization means that the patient can either be randomized to intervention (Evira Care) or control (Standard Lifestyle Care) group.

The study duration is 12 months. The Intervention group will receive Evira support (Evira Care) in combination with local standard treatment (Standard Lifestyle Care). During the first 2-4 weeks, they will receive information about the system and how to utilize the daily weighings and communication system. The families will be informed about possible lifestyle changes that may be effective. Furthermore, they will be informed that they are supposed to do lifestyle changes primarily regarding energy intake that they do consider feasible in their specific living situations. Within four weeks after randomization, the families will get one or two scales, depending on the family situation. The parent's will also have the mobile app installed in their smart phones and, depending on the age of the child, in the child's phone as well. The individual weight loss target curve for the first three months of treatment will be installed in the database and presented in the application. The control group will receive Standard Lifestyle Care without any restriction in visits or clinical support.

The following clinical investigations will be completed in both groups: 1) Physical examination including puberty, cardio-respiratory, thyroid status, skin (e.g. acanthosis nigricans) and abdominal examinations, and 2) Weight, height, and blood pressure. Blood sampling in accordance with local routine can be reported at any time-point.

In addition to the clinical investigation, all participants will be asked to answer questionnaires including quality of life, eating disorders, and treatment satisfaction. Background information and negative side effects will be reported in the electronic case report form (e-crf).

ELIGIBILITY:
Inclusion Criteria:

* Age >4.0 and <17.0 years of age at inclusion
* Obesity defined based on the International Obesity Task Force criteria iso-BMI 30 - 40 kg/m2
* Willingness to participate in an obesity treatment clinical trial
* Family ability to communicate in the language of the country of residence e.g. write and read messages in the mobile application
* Parents having a smart phone and an email address

Exclusion Criteria:

* Morbid obesity defined as iso-BMI>40kg/m2 independently of age
* Endocrine disorders other than well controlled hypothyroidism
* Metabolic disorders of importance for weight control - to be discussed
* Treatment for depression and other psychiatric disorders during the last 6 months before inclusion
* Pharmacological treatment of importance for weight control
* Hypothalamic or monogenic obesity, e.g. syndromes and Mb Down
* Severe neuropsychiatric disorders that could affect study compliance
* Eating disorders requiring therapy during the last six months before inclusion or observed at the inclusion screening.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 680 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in degree of obesity | Baseline, 12-month follow-up
  Measured by BMI standard deviation score. Support system users vs. control

SECONDARY OUTCOMES:
Treatment compliance | Baseline, 12-month follow-up
  Measured by number of physical visits, cancellations, Evira weighings, communication through the system and no-shows
Psycho-social health measures | Baseline, 12-month follow-up
  Psycho-social health assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire. The PROMIS questionnaire is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. The output from a PROMIS score is represented as a T-score. Higher scores indicate more of the domain being measured (e.g., more fatigue, more pain).

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Danielsson, PhD, Principal Investigator — Karolinska Institutet
Locations (5):
- Italy (2):
  - University of Messina, Messina
  - University of Campania Luigi Vanvitelli, Naples
- St. Olavs Hospital, Trondheim, Norway
- Samodzielny Publiczny Szpital Kliniczny, Szczecin, Poland
- Kalmar barnklinik, Kalmar, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data for the main outcome will be available upon date of scientific publications. To preserve individual case and anonymity, more detailed data and additional variables will be available upon request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will become available upon date of scientific publications or on requests.